CLINICAL TRIAL: NCT06838039
Title: Assessing the Impact of Additional Serratus Anterior Block Within 24-Hour on Postoperative Pain After Rhomboid Intercostal Block in VATS Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Quds University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Re27-06-024
Record Dates: First submitted 2025-01-20; First posted 2025-02-20 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Pain; VATS
Keywords: Postoperative Pain Management; Video-Assisted Thoracoscopic Surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (RIB Only) (Experimental): Participants receive a Rhomboid Intercostal Block (RIB) as the sole regional anesthesia technique for postoperative pain management after VATS
  Interventions: Procedure: Rhomboid Intercostal Block (RIB)
- Arm 2 (RIB + SAPB) (Experimental): Participants receive both RIB and SAPB within 24 hours postoperatively
  Interventions: Procedure: Rhomboid Intercostal Block (RIB) + Serratus Anterior Plane Block (SAPB)

INTERVENTIONS:
Procedure: Rhomboid Intercostal Block (RIB) — Rhomboid Intercostal Block (RIB) A regional anesthesia technique administered under ultrasound guidance for postoperative pain relief. This will be used as the sole intervention in Arm 1.
  Arms: Arm 1 (RIB Only)
Procedure: Rhomboid Intercostal Block (RIB) + Serratus Anterior Plane Block (SAPB) — A combination of two regional anesthesia techniques, Rhomboid Intercostal Block (RIB) and Serratus Anterior Plane Block (SAPB),(THE SAPB will received within 24 hours after RIB) administered under ultrasound guidance. SAPB targets the lateral cutaneous branches of the thoracic nerves, complementing the pain relief provided by RIB. This combination is used in Arm 2 to enhance postoperative analgesia.
  Arms: Arm 2 (RIB + SAPB)

SUMMARY:
Title: Assessing the Impact of Additional Serratus Anterior Block on Postoperative Pain After Rhomboid Intercostal Block in VATS Patients

Purpose: This randomized controlled trial aims to evaluate whether the addition of a Serratus Anterior Plane Block (SAPB) to the standard Rhomboid Intercostal Block (RIB) improves postoperative pain management in patients undergoing Video-Assisted Thoracoscopic Surgery (VATS).

Study Design:

* Type: Randomized Controlled Trial (RCT)
* Participants: 50 patients aged 18 -70 requiring VATS, randomized into two groups: one receiving RIB alone, and the other receiving RIB + SAPB.
* Duration: Pain and opioid consumption will be measured within 48 hours post-surgery.
* Outcome Measures: Pain levels using the Visual Analog Scale (VAS), opioid usage, and patient satisfaction.

Significance:

The study addresses the gap in research regarding the combined use of SAPB and RIB in pain control for VATS. It hypothesizes that the combination will lead to better pain relief and reduced opioid dependence compared to RIB alone.

DETAILED DESCRIPTION:
Title: Assessing the Impact of Additional Serratus Anterior Plane Block on Postoperative Pain After Rhomboid Intercostal Block in VATS Patients

Background:

Video-Assisted Thoracoscopic Surgery (VATS) is a minimally invasive thoracic procedure that has revolutionized the treatment of lung diseases, pleural conditions, and mediastinal disorders. While it offers numerous advantages, including smaller incisions, shorter hospital stays, and faster recovery, postoperative pain remains a significant challenge. Uncontrolled pain can impair pulmonary function, delay ambulation, and increase the need for opioids, which in turn elevates the risk of opioid-related side effects such as respiratory depression, nausea, and addiction potential.

Regional anesthesia techniques, particularly Rhomboid Intercostal Block (RIB), have gained popularity as effective methods for postoperative pain control following VATS. RIB is an ultrasound-guided technique that targets the intercostal nerves by depositing local anesthetic into the fascial plane between the rhomboid and intercostal muscles. This block has demonstrated efficacy in reducing pain intensity and opioid consumption in VATS patients. However, some patients may still experience inadequate pain relief, particularly in areas not covered by RIB alone.

The Serratus Anterior Plane Block (SAPB) is another regional anesthesia technique that anesthetizes the lateral cutaneous branches of the thoracic intercostal nerves, which contribute to the sensory innervation of the chest wall. Given that SAPB and RIB target different pain pathways, combining these two blocks may provide broader and more effective analgesia for VATS patients.

While SAPB has been successfully utilized in thoracic surgeries, limited data exist regarding its additive effect when used in conjunction with RIB. This study aims to evaluate whether SAPB, when administered within 24 hours after RIB, provides superior postoperative pain control compared to RIB alone.

Scientific Rationale:

Postoperative pain in VATS originates from multiple sources, including surgical incision sites, pleural irritation, and muscle disruption. The intercostal nerves supply the majority of sensory innervation to the chest wall, making them primary targets for regional anesthesia.

* RIB blocks the dorsal rami of intercostal nerves, leading to effective posterior thoracic analgesia. However, it may not completely cover the lateral and anterior chest wall, which are innervated by lateral cutaneous branches.
* SAPB, on the other hand, targets the lateral cutaneous branches of the intercostal nerves, complementing the analgesia provided by RIB and potentially enhancing the overall pain relief.

By combining RIB and SAPB, this study hypothesizes that patients will experience superior pain relief, reduced opioid consumption, and improved satisfaction compared to RIB alone. This multimodal approach aligns with the growing emphasis on opioid-sparing anesthesia strategies.

Study Objective:

The primary objective of this randomized controlled trial is to evaluate whether the addition of SAPB to standard RIB improves postoperative pain control, reduces opioid consumption, and enhances patient satisfaction within 48 hours after VATS surgery.

Methodology

* Study Design: A prospective, randomized controlled trial.
* Participants: Adult patients (ages 18-70) undergoing VATS surgery.
* Group Allocation:
* Group A (Control Group): RIB only.
* Group B (Intervention Group): RIB + SAPB (SAPB administered within 24 hours after RIB).
* Primary Outcome Measure:
* Pain severity assessed using the Visual Analog Scale (VAS) at multiple postoperative time points.
* Secondary Outcome Measures:
* Total opioid consumption within 48 hours.
* Patient satisfaction scores via standardized questionnaires.
* Incidence of complications or adverse effects related to regional anesthesia.
* Blinding: The outcome assessor will be blinded to the intervention groups to reduce bias.
* Data Collection and Analysis:
* Baseline demographic and clinical data will be recorded.
* Statistical analysis will compare pain scores, opioid use, and satisfaction levels between the two groups.
* Subgroup analyses may be performed based on VATS procedure types or patient demographics.

Expected Outcomes

We hypothesize that the combination of SAPB with RIB will result in:

* Significant reductions in pain scores within 48 hours.
* Lower opioid consumption compared to RIB alone.
* Higher overall patient satisfaction with pain management. If successful, this study could provide strong clinical evidence supporting the routine use of SAPB alongside RIB for VATS pain control.

Significance:

This study addresses an important gap in postoperative pain management for VATS patients. While RIB alone is widely used, its efficacy in providing complete analgesia is still under debate. By exploring the synergistic effects of SAPB and RIB, this trial aims to advance regional anesthesia techniques and contribute to more effective, multimodal pain management strategies.

The results of this study have potential clinical implications for thoracic anesthesia practice, particularly in settings where minimizing opioid use is a priority due to concerns about addiction, side effects, and prolonged hospital stays.

Trial Locations:

The trial will be conducted at Al-Ahli and Al-St. Joseph's Hospitals, Palestine, where VATS procedures are routinely performed.

Budget and Resource Allocation

* Participant recruitment and informed consent process.
* Materials for data collection, including VAS scales and patient satisfaction questionnaires.
* Statistical analysis software to ensure robust data interpretation.
* Ultrasound guidance equipment and anesthetic agents for RIB and SAPB administration

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-70 years.
2. Patients undergoing Video-Assisted Thoracoscopic Surgery (VATS).
3. Classified as ASA physical status I-III (low to moderate surgical risk).
4. Ability to provide informed consent and follow study protocols.

Exclusion Criteria:

1. Known allergy or hypersensitivity to local anesthetics.
2. Presence of bleeding disorders or anticoagulant use.
3. History of chronic opioid use or opioid dependence.
4. Anatomical abnormalities or conditions preventing the application of regional anesthesia (e.g., chest wall deformities).
5. Presence of neurological disorders affecting pain perception.
6. Cognitive impairments, language barriers, or inability to communicate effectively.
7. Pregnancy or breastfeeding.
8. Refusal or inability to provide informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain Severity | 48 hours post-surgery.
  Postoperative pain will be assessed using the Visual Analog Scale for pain which higher score mean more pain at various time intervals (e.g., 1,12, 24, 36 and 48 hours post-surgery).

SECONDARY OUTCOMES:
Opioid Consumption | 48 hours post-surgery.
  Total opioid consumption (measured in morphine milligram equivalents) during the first 48hours post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Al Ahli hospital, Hebron, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No